CLINICAL TRIAL: NCT04571853
Title: Usefulness of a New Educational Tool for Understanding Pain for Fibromyalgia Patients
Brief Title: New Educational Tool for FM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: University of South Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEW EDUCATION TOOL
Record Dates: First submitted 2020-09-26; First posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Pain Neuroscience Education; Pain; Fact Sheets
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Single-blind, parallel-group, randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PNE-explained group (Experimental): The participants in the PNE-explained group will be explained the fact sheets with an explanatory video (due to COVID-19 circumstances) conducted by the therapist M.S. The video will last one hour approximately and it contains a presentation by Mayte Serrat with a view of the fact sheets. This group will be given one week to watch the video and comprehend its content.
  Interventions: Behavioral: PNE-explained group
- PNE-read group (Active Comparator): The PNE-read group will receive the fact sheets via email along with instructions regarding the content and the procedure to read the content. Instructions will suggest to read only two fact sheets per day during 4,5 days. It will be suggested to take 30 minutes at least for each fact sheet.
  Interventions: Behavioral: PNE-read group
- TAU group (Active Comparator): Participants allocated into this group will maintain treatment as usual (TAU) and will follow the recommendations by their usual health professional.
  Interventions: Behavioral: TAU group

INTERVENTIONS:
Behavioral: PNE-explained group — There are 9 fact sheets overall. And each fact sheet incorporates two pages relating to one main concept. The first of two pages introduces the concept, and the second one quotes important ideas that emerge from the main concept. The 9 main concepts and consequent ideas presented in the fact sheets are based on current scientific research in pain science and have been selected and structured specifically for PNE education for chronic pain patients. The fact sheets have been fully developed and designed by Pain Revolution, a pain educator network founded by Professor Lorimer Moseley, group leader in Body in Mind Research Group from University of South Australia.
  Arms: PNE-explained group
Behavioral: PNE-read group — The PNE-read group will receive the fact sheets via email along with instructions regarding the content and the procedure to read the content. Instructions will suggest to read only two fact sheets per day during 4,5 days. It will be suggested to take 30 minutes at least for each fact sheet.
  Arms: PNE-read group
Behavioral: TAU group — Participants allocated to this group will maintain treatment as usual (TAU) and will follow the recommendations by their usual health professiona
  Arms: TAU group

SUMMARY:
This study aims at analyzing the usefulness of a new educational tool developed by Pain Revolution, a compendium of 9 fact sheets along with a related quiz in patients from the Hospital Vall d'Hebron of Barcelona suffering from fibromyalgia, compared to a non-education group. The present study also aims at comparing the usefulness of the new tool based on PNE in two different formats: read and explained.

DETAILED DESCRIPTION:
Main objective

A compendium of 9 fact sheets along with a related quiz have been developed in order to provide overall population current pain-science knowledge. The present study aims at analyzing the usefulness of this new tool based on pain neuroscience education (PNE) in patients from the Hospital Vall d'Hebron of Barcelona suffering from fibromyalgia, compared to a non-education group.

Secondary objective

Due to the extended content of the fact sheets, these can be delivered to the patient as a reading material or can be used as a support material in a educational presentation. Therefore, this study also aims at comparing the usefulness of the new tool based on PNE in two different formats: read autonomously by the patient and explained by a pain-science expert to the patient.

This is a tree-arm RCT: TAU group and intervention group with 2 different groups as follows:

The intervention program is divided in two groups. Both groups will be provided with the PNE fact sheets but in different format (read and explained) and will be given one week to comprehend the content before to assess their knowledge. Therefore, intervention groups will be informed that a quiz about the fact sheets will be delivered to each one in order to asses their acquired knowledge.

There are 9 fact sheets overall. And each fact sheet incorporates two pages relating to one main concept. The first of two pages introduces the concept, and the second one quotes important ideas that emerge from the main concept. The 9 main concepts and consequent ideas presented in the fact sheets are based on current scientific research in pain science and have been selected and structured specifically for PNE education for chronic pain patients. The fact sheets have been fully developed and designed by Pain Revolution, a pain educator network founded by Professor Lorimer Moseley, group leader in Body in Mind Research Group from University of South Australia.

ELIGIBILITY:
Inclusion Criteria:

* Adults from 18 to 75 years-old.
* 1990 American College of Rheumatology (ACR) classification criteria + the 2011 modified ACR diagnostic criteria for fibromyalgia
* Able to understand Spanish and accept to participate in the study.

Exclusion Criteria:

* Participating in concurrent or past RCTs (previous year).
* Comorbidity with severe mental disorders (i.e. psychosis) or neurodegenerative diseases (i.e. Alzheimer) that that would limit the ability of the patient to participate in the RCT.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-10-10 (Estimated); Study Completion 2021-10-10 (Estimated)

PRIMARY OUTCOMES:
Pain Revolution Quiz | Through study completion, an average of 1 week]
  The Pain Revolution Quiz comprises two main sections: one first section related to the acquired knowledge after the fact sheets and the second section incorporates 4 questions with feedback about the learning process. The first section encompasses 26 items which are used to measure acquired knowledge by the subjects after being provided the 9 fact sheets content. The 26 items are answered on multicomponent choices of three possible alternatives: true, false and I don't know. Total scores can range from 0 to 26. Some of the items respond to reverse score, such as 1, 5, 7, 8, 10, 12, 14, 20, 22, 25, 26. This tool has been recently developed by Pain Revolution, a pain educator network founded by Professor Lorimer Moseley, group leader in Body in Mind Research Group from University of South Australia. The adequate internal consistency and acceptable test-retest reliability is currently being studied. In the same manner, the Spanish version is evaluated for first time in the present study.

CONTACTS AND LOCATIONS:
Overall Officials: Lorimer Moseley, PhD, Principal Investigator — University of South Australia; Sara Marsall, PhD, Study Director — Hospital Universitari Vall dHebron
Locations (1):
- Mayte Serrat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No